CLINICAL TRIAL: NCT03648775
Title: National, Multicentre, Prospective, Observational Study, to Evaluate the Clinical Efficacy of Y-STRUT® Medical Device Implanted for Contralateral Percutaneous Internal Fixation of Proximal Femur, in Patient With a Low Energy Per Trochanteric Fracture on the First Side
Brief Title: Evaluation of the Clinical Efficacy of Y-STRUT® Medical Device Implanted for Contralateral Percutaneous Internal Fixation of Proximal Femur, in Patient With a Low Energy Per Trochanteric Fracture on the First Side
Status: Terminated | Type: Observational
Why Stopped: Suspension of the study upon the decision of the notified body
Sponsor: Hyprevention (Industry)
Responsible Party: Sponsor
Other Study IDs: HIP50
Record Dates: First submitted 2018-08-21; First posted 2018-08-27 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Fracture of Hip; Osteoporosis
Keywords: Osteosynthesis; Prophylactic consolidation; Proximal femur
MeSH Terms: conditions — Hip Fractures; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Y-STRUT® (Hyprevention, Pessac, France) — The studied medical device consists of two components implanted in the proximal femur, combined with bone cement.

SUMMARY:
HIP50 is a national, multicentre, prospective, observational study, in patients presenting a first low energy per trochanteric hip fracture on one side and treated with Y-STRUT® device implanted on the contralateral proximal femur as percutaneous internal fixation to prevent contralateral hip fracture in case of osteoporosis.

The primary objective of this study is to evaluate the clinical efficacy of the studied medical device by measuring the frequency of patient with a fracture at the implantation site within 1 year after implantation.

A total of 50 patients from France will be enrolled (until December 2020) and followed up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient of 60 years and older, according to CE indication;
* Patient with information form signed to participate in the study;
* Patients presenting a first low energy hip fracture on one side and having a Y-STRUT® device implanted on the contralateral hip between 0 and 120 days after the treatment of the fracture of the first hip;

Exclusion Criteria:

* Patient who refuse to participate to this study;
* Patient implanted with Y-STRUT® for another indication;
* Patient already enrolled in a clinical study, excluding his participation to HIP50.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting a first low energy per trochanteric hip fracture on one side and treated with Y-STRUT® device implanted on the contralateral proximal femur as percutaneous internal fixation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Frequency of post-operative fracture [Clinical efficacy of the device] | At 12 months
  Frequency of Y-STRUT® implanted patients with a fracture at the implantation site

SECONDARY OUTCOMES:
Frequency of post-operative fracture [Clinical efficacy of the device] | At 3 and 24 months
  Frequency of Y-STRUT® implanted patients with a fracture at the implantation site
Recording of concomitants treatments [safety and feasibility of the device] | At 3, 12 and 24 months
  Recording of all concomitants treatments: analgesic for pain, anti-osteoporotic treatment and other treatments.
Pain [safety and feasibility of the device] | At 3, 12 and 24 months
  Self-evaluation of hip pain using VAS (Visual Analogue Scale), going from 0 (no pain) to 10 (maximum).
Walking conditions [safety and feasibility of the device] | At 3, 12 and 24 months
  Assessment of resumption of weight-bearing (yes/no, aid)
Recording of adverse events and device effects [safety and feasibility of the device] | At 3, 12 and 24 months
  Recording of the medical device vigilance: all serious adverse events, all adverse events linked to the device or the operative technique, and any other important event reported.
Surgical procedure duration [learning curve of the procedure] | At the end of the inclusion period (24 months from the first included patient)
  Measuring mean/median intervention duration of each procedure. Then, all the durations of successive procedures will be compared among all the investigators.
Hospitalisation duration [learning curve of the procedure] | At the end of the inclusion period (24 months from the first included patient)]
  Measuring mean/median hospitalisation duration. Then, all the durations of successive hospitalisations will be compared among all the investigators.
Rate of complications [learning curve of the procedure] | At the end of the inclusion period (24 months from the first included patient)
  Assessing types and frequencies of procedures complications (per-op and post-op). Then, all the rate of complications will be compared among all the investigators.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Hôpital Privé d'Ambérieu, Ambérieu-en-Bugey
  - Hôpital Antoine Béclère, Clamart
  - Centre Hospitalier Universitaire Grenoble Alpes, La Tronche
  - Centre Hospitalier Régional Orléans, Orléans
  - Nouvelle Clinique de Tours Plus St Gatien, Tours